CLINICAL TRIAL: NCT01027052
Title: Absorption, Metabolism and Antioxidant Effects of Common Herbs
Brief Title: Spices Inhibit the Formation and Absorption of Malondialdehyde From Hamburger Meat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 08-03-008-01
Record Dates: First submitted 2009-08-13; First posted 2009-12-07 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: NIDDM
Keywords: MDA; Spice
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Salts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hamburger meat patty with Spice Blend (Active Comparator): Hamburger meat patty containing spice blend will be consumed on 3 separate occasions
  Interventions: Other: Hamburger meat patty with spice blend
- Hamburger meat patty with salt (Placebo Comparator): Hamburger meat patty containing salt will be consumed on 3 separate occasions
  Interventions: Other: Hamburger meat patty with salt

INTERVENTIONS:
Other: Hamburger meat patty with salt — hamburger meat cooked with salt
  Arms: Hamburger meat patty with salt
Other: Hamburger meat patty with spice blend — hamburger meat cooked with spice mixture
  Arms: Hamburger meat patty with Spice Blend

SUMMARY:
Polyphenols belong to the largest group of secondary metabolites produced by plants, mainly, in response to biotic or abiotic stresses such as infections, wounding, UV irradiation, exposure to ozone, pollutants, and other hostile environmental conditions. It is thought that the molecular basis for the protective action of polyphenols in plants is their antioxidant and free radical scavenging properties. These numerous phenolic compounds are major biologically active components of spices, aromas, essential oils, and traditional medicines. In order to investigate the impact of spice polyphenols on postprandial cytotoxic lipid peroxidation products (MDA) levels in humans, the investigators propose to achieve the following specific aims using a randomized crossover study design:

1. To determine the effect of a ground beef patty meal with and without spices on postprandial levels of plasma malondialdehyde (MDA).
2. To determine the effect of a ground beef patty meal with and without a spice blend on MDA accumulation in urine.

This study will determine whether spice polyphenols exert a beneficial effect by inhibition of the absorption of MDA. These findings may help to explain the potentially harmful effects of oxidizable fats found in foods and the important benefit of dietary polyphenols in ameliorating this potentially harmful effect.

DETAILED DESCRIPTION:
10 male subjects with type 2 diabetes mellitus who will be recruited based on inclusion and exclusion criteria. The study will be carried out in accordance with the guidelines of the Human Subjects Protection Committee of the University of California, Los Angeles. All subjects will give written informed consent before the study begins. After the screening visit, each subject will come to the Center for Human Nutrition on two 1-day test phases separated by at least one week. At each of phases, subjects will consume, in a random order, two different test meals consisting of either: a) a ground dark meat beef patty seasoned with salt only, or b) a ground dark meat beef patty seasoned with a spice mixture and salt. The subjects will be asked to avoid eating meat, poultry, or fish products for 3 days before the day of each of the two experimental phases

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 20-45 years of age
* Non-smokers, or smoke < 1 cigarette per day
* Not exercising heavily (< 4 x 30 minutes aerobic exercise per week)
* Willing to maintain normal activity and eating patterns for the duration of the study
* Willing to avoid meat, fish or poultry for three days on two occasions prior to the test procedure
* Consuming less than two alcoholic drinks per day
* Not taking dietary supplements
* No known allergy to beef, cloves, cinnamon, oregano, turmeric, cumin, rosemary, sage, red pepper, ginger, black pepper, paprika or garlic

Exclusion Criteria:

* Metabolic disorders
* Taking dietary supplements
* Smoking >1 cigarette/day
* Exercising heavily (>4x30 min of aerobic exercise/wk)
* Drinking more than 2 glasses of wine, 2 cocktails or two beers /day.
* Allergic to beef, cloves, cinnamon, oregano, turmeric, cumin, rosemary, sage, red pepper, ginger, black pepper, paprika or garlic
* Known HIV positive

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Change in plasma and urinary MDA after consumption of hamburg with or without spice mixture added | 2 days
  Change in plasma and urinary MDA after consumption of 250 g hamburg meat with 11.3 g spice mixture added or without spice

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — David Geffen School of Medicine, UCLA Center for Human Nutrtiion

REFERENCES:
- [Derived] Li Z, Henning SM, Zhang Y, Zerlin A, Li L, Gao K, Lee RP, Karp H, Thames G, Bowerman S, Heber D. Antioxidant-rich spice added to hamburger meat during cooking results in reduced meat, plasma, and urine malondialdehyde concentrations. Am J Clin Nutr. 2010 May;91(5):1180-4. doi: 10.3945/ajcn.2009.28526. Epub 2010 Mar 24. PMID 20335545